CLINICAL TRIAL: NCT05275491
Title: Serum Levels of Fibroblast Growth Factor 23 and Sclerostin in Relation to Serum Calcium Level in COVID 19 Patients
Brief Title: Fibroblast Growth Factor 23 and Sclerostin in Relation to Calcium in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Asmaa Abdel-mageed Muhammed, Lecturer, Aswan University Hospital
Other Study IDs: FGF23 in COVID-19
Record Dates: First submitted 2022-03-10; First posted 2022-03-11 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19; Hypocalcemia; Fibroblast growth factor 23 (FGF23); Sclerostin
MeSH Terms: conditions — COVID-19; Hypocalcemia; Sclerosteosis | interventions — Calcium Signaling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild to moderate COVID 19 patients: According to COVID 19 treatment guidelines of National Institutes of Health (NIH):
  Mild illness that show symptoms like fever, cough, nausea, vomiting, sore throat, loss of taste & smell but don't show dyspnea or abnormal chest imaging.
  Moderate illness that show clinical or radiological lower respiratory disease with SpO2 > 94% on room air.
  Interventions: Diagnostic Test: Calcium; Diagnostic Test: Fibroblast growth factor 23; Diagnostic Test: Sclerostin; Diagnostic Test: parathyroid hormone
- Severe to critical COVID 19 patients: According to COVID 19 treatment guidelines of National Institutes of Health (NIH):
  Severe illness that show SpO2 < 94% on room air, (PaO2/FiO2) <300 mm Hg & lung infiltration > 50% with respiratory rate > 30 breath/min.
  Critical illness that show respiratory failure, septic shock or multiorgan failure.
  Interventions: Diagnostic Test: Calcium; Diagnostic Test: Fibroblast growth factor 23; Diagnostic Test: Sclerostin; Diagnostic Test: parathyroid hormone
- Normal male subjects (Control)
  Interventions: Diagnostic Test: Calcium; Diagnostic Test: Fibroblast growth factor 23; Diagnostic Test: Sclerostin; Diagnostic Test: parathyroid hormone

INTERVENTIONS:
Diagnostic Test: Calcium — Free calcium serum levels
Diagnostic Test: Fibroblast growth factor 23 — Serum level
Diagnostic Test: Sclerostin — Serum level
Diagnostic Test: parathyroid hormone — serum level

SUMMARY:
Hypocalcemia is associated with COVID-19 patients and is linked to poor prognosis, Fibroblast growth factor 23 (FGF23) and Sclerostin inhibit vitamin D activation and are linked to hypocalcemia.

Levels of FGF23 and Sclerostin in COVID-19 patients will be detected and correlated to calcium levels.

DETAILED DESCRIPTION:
COVID 19 is a current worldwide pandemic caused by severe acute respiratory syndrome coronavirus 2 "SARS-CoV-2". Hypovitaminosis D and hypocalcaemia have been reported to be associated with COVID 19 infection, they are considered good biomarkers of clinical severity of COVID 19. Poor prognosis related to hypocalcemia is increased in elderly patients.

Fibroblast growth factor 23 and sclerostin are secreted from the bone, they decrease active vitamin D levels. Their levels and their relation to calcium levels in COVID-19 patients will be detected.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID 19 (Mild to moderate - severe to critical).

Exclusion Criteria:

* known diagnosis of CKD.
* Known parathyroid disease.
* Use of phosphate binder therapy within the past 3 months.
* Use of calcium therapy within the past 3 months
* Treatment with 25(OH) vitamin D or 1,25 (OH)(2) D
* Underlying metabolic bone disease.
* Underlying renal phosphate wasting disorder.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (Group A): Mild to moderate COVID 19 patients. (Group B): Severe to critical COVID 19 patients. (Group C): Normal male subjects (Control)
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in serum calcium levels | 6 months
  Expected lower serum calcium levels in COVID 19 patients compared to control
changes in FGF23 levels | 6 months
  Expected higher FGF23 levels in COVID 19 patients compared to control
changes in sclerostin levels | 6 months
  Expected higher sclerostin levels in COVID 19 patients compared to control
Changes in parathyroid hormone levels | 6 months
  Expected lower levels in COVID 19 patients compared to control

SECONDARY OUTCOMES:
Relation between FGF 23 and calcium levels | 6 months
  A negative relation is expected
Relation between sclerostin and calcium levels | 6 months
  A negative relation is expected

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Abdelmageed Muhammed, Lecturer, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University hospital, Aswān, Egypt

REFERENCES:
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Background] Zhou X, Chen D, Wang L, Zhao Y, Wei L, Chen Z, Yang B. Low serum calcium: a new, important indicator of COVID-19 patients from mild/moderate to severe/critical. Biosci Rep. 2020 Nov 30;40(12):BSR20202690. doi: 10.1042/BSR20202690. Online ahead of print. PMID 33252122
- [Background] Demir M, Demir F, Aygun H. Vitamin D deficiency is associated with COVID-19 positivity and severity of the disease. J Med Virol. 2021 May;93(5):2992-2999. doi: 10.1002/jmv.26832. Epub 2021 Feb 9. PMID 33512007
- [Background] di Filippo L, Doga M, Frara S, Giustina A. Hypocalcemia in COVID-19: Prevalence, clinical significance and therapeutic implications. Rev Endocr Metab Disord. 2022 Apr;23(2):299-308. doi: 10.1007/s11154-021-09655-z. Epub 2021 Apr 13. PMID 33846867
- [Background] Lewiecki EM. Role of sclerostin in bone and cartilage and its potential as a therapeutic target in bone diseases. Ther Adv Musculoskelet Dis. 2014 Apr;6(2):48-57. doi: 10.1177/1759720X13510479. PMID 24688605
- [Background] Quarles LD. Role of FGF23 in vitamin D and phosphate metabolism: implications in chronic kidney disease. Exp Cell Res. 2012 May 15;318(9):1040-8. doi: 10.1016/j.yexcr.2012.02.027. Epub 2012 Mar 7. PMID 22421513